CLINICAL TRIAL: NCT05698823
Title: Regular Home-use of Dual-light Photodynamic Therapy in the Management of Chronic Stage III-IV Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: University of Helsinki (Other); Lithuanian University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LumoKaunas2023
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis Chronic Generalized Moderate; Periodontitis Chronic Generalized Severe
Keywords: Lumoral; Lumorinse; Periodontitis; Anti-bacterial photodynamic therapy; aPDT; Plaque; aMMP-8; Photobiomodulation
MeSH Terms: conditions — Periodontitis; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All clinical assessments at baseline and at 6 months shall be performed by one calibrated examiner who is blinded for the subjects' allocation to the study and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): A complete clinical intraoral examination shall be performed for all subjects. Same demographic and clinical data will be obtained from subjects in both arms. The study group shall receive the Lumoral treatment -device, Lumorinse -tablets and instructions for their use.
  All subjects shall receive standard oral hygiene instructions for the use of an electric toothbrush, interdental brush, and dental floss.
  Interventions: Device: Lumoral Treatment
- Control group (No Intervention): A complete clinical intraoral examination shall be performed for all subjects. Same demographic and clinical data will be obtained from subjects in both arms. All subjects shall receive standard oral hygiene instructions for the use of an electric toothbrush, interdental brush, and dental floss.

INTERVENTIONS:
Device: Lumoral Treatment — The Lumoral treatment -device is a CE-marked antibacterial home-use device for the treatment and prevention of oral diseases caused by bacteria. It is used in combination with a CE-marked mouth rinse called Lumorinse.
  Arms: Study group

SUMMARY:
This study is designed to determine the efficacy of the Lumoral method in chronic periodontitis with a targeted group of stage III and IV periodontitis.

Improved supragingival plaque control can help to also sustain the subgingival plaque management in the long term.

In addition, the method might have a photobiomodulation effect on periodontal tissues.

DETAILED DESCRIPTION:
The Lumoral Treatment is a CE-marked medical device developed to provide a potent, targeted antibacterial action on dental plaque in a home environment. The device mechanism of action is antibacterial photodynamic therapy (aPDT). The device is used by swishing a specially designed mouth rinse that strongly adheres to dental plaque. The plaque-adhered photoactive mouth rinse can be activated by a simple-to-use light applicator. Preliminary results have shown promising anti-inflammatory responses in addition to plaque reduction.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal disease stage III-IV, according to criteria the American Academy of Periodontology (AAP) with at least 3 mm interdental clinical attachment level (CAL) in the site of greatest loss.
* ≥ 18 years old
* Presence of ≥20 teeth, including implants
* Agreement to participate in the study and to sign a written consent form
* Able to co-operate with the treatment protocol and avoid any other oral hygiene measures outside of the study protocol

Exclusion Criteria:

* Grade A or C periodontitis
* Presence of any physical limitation or restriction that might restrict Lumoral use
* Pregnancy or lactation
* Active smoking
* Medicated diabetes mellitus (DM)
* Any systemic disease (e.g., wound healing dysfunctions) that could alter the progression of periodontal disease
* Use of antibiotics within 4 weeks week prior study
* Periodontal treatment within 3 months prior study
* Removable major prosthesis or major orthodontic appliance
* A need for a hopeless teeth extraction, or open cavities in need for immediate endodontic treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) | 6 months
  Improvement in bleeding on probing (BOP)
  * A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual)
  * Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus
  * Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent"
  * BOP is reported as the percentage (%) of sites with positive findings
  * Calculation formula: number of bleeding sites/ 6 times number of teeth

SECONDARY OUTCOMES:
Active matrix metalloproteinase 8 (aMMP-8) | 6 months
  Change in periodontal inflammation marker aMMP-8
Visible plaque index (VPI) | 6 months
  Change in visible plaque index (VPI)
Probing pocket depth (PPD) | 6 months
  Change in probing pocket depth (PPD)
Clinical attachment level (CAL) | 6 months
  Change in clinical attachment level (CAL)
Deep periodontal pockets (over 4 mm) | 6 months
  Change in the number of deep periodontal periodontal pockets (over 4 mm)
Periodontal microbiological flora | 6 months
  Change in periodontal microbiological flora during the study period
Additional visits | 6 months
  Number of additional visits due to periodontitis status between 2nd and 3rd follow-up visits
OHIP-14 | 6 months
  Patient related objectives: Oral-related quality of life measurement (OHIP-14) questionnaire

OTHER OUTCOMES:
Device-related adverse event | 6 months
  Absence of device-related serious adverse events or any patterns of device-related adverse events graded as moderate

CONTACTS AND LOCATIONS:
Overall Officials: Timo Sorsa, Professor, Study Director — University of Helsinki; Tommi Pätilä, Docent, Study Chair — Koite Health; Ingrida Marija Pacauskiene, Doctor, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Department of Dental and Oral Pathology, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No
The IPD will only be administered by the researchers that are listed in the CIP.

REFERENCES:
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of severe periodontitis in 1990-2010: a systematic review and meta-regression. J Dent Res. 2014 Nov;93(11):1045-53. doi: 10.1177/0022034514552491. Epub 2014 Sep 26. PMID 25261053
- [Background] Kassebaum NJ, Smith AGC, Bernabe E, Fleming TD, Reynolds AE, Vos T, Murray CJL, Marcenes W; GBD 2015 Oral Health Collaborators. Global, Regional, and National Prevalence, Incidence, and Disability-Adjusted Life Years for Oral Conditions for 195 Countries, 1990-2015: A Systematic Analysis for the Global Burden of Diseases, Injuries, and Risk Factors. J Dent Res. 2017 Apr;96(4):380-387. doi: 10.1177/0022034517693566. PMID 28792274
- [Background] Lang NP, Suvan JE, Tonetti MS. Risk factor assessment tools for the prevention of periodontitis progression a systematic review. J Clin Periodontol. 2015 Apr;42 Suppl 16:S59-70. doi: 10.1111/jcpe.12350. PMID 25496279
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- See also: Alaijah, F., Morsi, A., Nasher, R. et al. Photobiomodulation therapy in the treatment of periodontal disease: a literature review. Laser Dent Sci 3, 147-153 (2019) — https://doi.org/10.1007/s41547-019-00056-9
- See also: Gomes SC, Romagna R, Rossi V, Corvello PC, Melchiors-Angst PD. Supragingival treatment as an aid to reduce subgingival needs: a 450-day investigation Braz. oral res. 28 (1) 2014 — https://doi.org/10.1590/S1806-83242014.50000004
- See also: Levine JI. Medications that increase photosensititivity. FDA document Dec 1990. — https://www.fda.gov/media/75892/download
- See also: Nikinmaa S, Alapulli H, Auvinen P, et al. (2020) Dual-light photodynamic therapy administered daily provides a sustained antibacterial effect on biofilm and prevents Streptococcus mutans adaptation. PLoS ONE 15(5): e0232775 — https://doi.org/10.1371/journal.pone.0232775
- See also: Pereira PAB, Aho VTE, Paulin L, et al., (2017) Oral and nasal microbiota in Parkinson's disease. Parkinsonism and Related Disorders 38: 61-67 — http://dx.doi.org/10.1016/j.parkreldis.2017.02.026